CLINICAL TRIAL: NCT04327986
Title: A Phase I/II Study of the Immune Checkpoint Inhibitor M7824 and the Immunocytokine M9241 in Combination With Stereotactic Body Radiation Therapy (SBRT) in Adults With Advanced Pancreas Cancer
Brief Title: Immune Checkpoint Inhibitor M7824 and the Immunocytokine M9241 in Combination With Stereotactic Body Radiation Therapy (SBRT) in Adults With Advanced Pancreas Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study closed to accrual due to the worsening risk: benefit ratio for participants receiving bintrafusp alfa (M7824).
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Udo Rudloff, MD, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 200074; 20-C-0074
Record Dates: First submitted 2020-03-28; First posted 2020-03-31 (Actual); Results first posted 2022-05-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-04

CONDITIONS: Histologically or Cytologically Confirmed Pancreatic Cancer; Unresectable or Borderline Resectable Pancreatic Cancer; Pancreatic Neoplasms; Pancreatic Cancer; Metastatic Pancreatic Cancer
Keywords: Neoadjuvant therapy; Anti-Tumor Activity; Synergistic Anti-cancer Activity; Combining Immunotherapy and Radiation Therapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — bintrafusp alfa protein, human; NHS-IL12 immunocytokine; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 Phase 1A/Arm 1A (Experimental): De-escalating doses of NHS-IL12 (M9241) in combination with bintrafusp alfa (M7824)
  Interventions: Drug: M7824; Drug: M9241
- Cohort 2 Phase 1B/Arm 1B (Experimental): De-escalating doses of NHS-IL12 (M9241) in combination with bintrafusp alfa (M7824) and stereotactic body radiotherapy (SBRT)
  Interventions: Drug: M7824; Drug: M9241; Radiation: SBRT
- Phase II Cohort 3/Arm 2 (Experimental): Recommended phase 2 dose (RP2D) of bintrafusp alfa (M7824) and NHS-IL12 (M9241) in combination with stereotactic body radiotherapy (SBRT)
  Interventions: Drug: M7824; Drug: M9241; Radiation: SBRT

INTERVENTIONS:
Drug: M7824 — Intravenous (IV) on Days 1 and 15 of every cycle
  Other Names: bintrafusp alfa
Drug: M9241 — Subcutaneous injection on Day 1 of every cycle
  Other Names: NHS-IL12
Radiation: SBRT — Radiation therapy will be starting on Day 17 (+5 days) of Cycle 1 and continue for 5 consecutive business days.
  Other Names: Stereotactic body radiotherapy
  Arms: Cohort 2 Phase 1B/Arm 1B; Phase II Cohort 3/Arm 2

SUMMARY:
Background:

Fewer than 10 percent of people with pancreas cancer can have surgery. Surgery gives the best outcome. Radiation therapy is usually used to make surgery possible. But it does not work for most people. Adding immunotherapy might help.

Objective:

To find a safe combined dose of Bintrafusp Alfa (M7824), NHS-IL12 (M9241, and radiation and to see if it causes pancreas cancer tumors to shrink.

Eligibility:

People ages 18 and older who have pancreas cancer and cannot have curative surgery

Design:

Participants will be screened under protocol 01-C-0129 with:

Medical history

Physical exam

Heart, urine, and blood tests

Scans. For this, participants will lie in a machine that takes pictures of the body. They may receive a contrast agent by vein.

Possible tumor biopsy

Participants will take the study drugs either alone or with radiation. They will get M7824 by vein every 2 weeks. They will get M9241 injected under the skin every 4 weeks. Participants who get radiation will get it 5 days in a row the first month.

Participants will have visits every 2 weeks. They will repeat screening tests.

If participants tumors shrink, they will have surgery. If their whole tumor is removed, they will stop treatment. They will otherwise continue treatment as long as they can tolerate it and it is helping them.

Participants will have visits 1 week and 1 month after they stop treatment. Then they will be contacted by phone or email for life. If they stop treatment for a reason other than their disease getting worse, they will have scans every 12 weeks.

DETAILED DESCRIPTION:
Background:

* At time of diagnosis, fewer than 10% of newly diagnosed pancreatic cancer patients present with resectable disease (patients who can undergo surgery) and patients able to undergo a margin-negative surgical resection (R0) are reported to have the most favorable outcome.
* Locally advanced, non-metastatic pancreas cancer (LAPC) is observed in up to 30% of all pancreas cancer patients at time of diagnosis (including both borderline resectable and non-resectable disease).
* The primary goal of neoadjuvant therapy in LAPC is, among tumor control and extension of survival, the conversion to resectable disease achieving a R0 resection.
* Radiation therapy (RT) is commonly used as neoadjuvant treatment for LAPC.
* However, currently used RT neoadjuvant treatment regimens result in only about 40%-60% of patients with borderline resectable pancreas cancer to undergo surgical resection, in initially unresectable LAPC patient conversion are even lower, with only 7% - 19% able to undergo resection.
* Combining immunotherapy and radiation therapy could synergistically improve anti-cancer activity.
* Bintrafusp alfa (M7824) is a bifunctional fusion protein consisting of an anti-programmed death ligand 1 (PD-L1) antibody functioning as an immune checkpoint inhibitor and the extracellular domain of transforming growth factor beta (TGF-beta) receptor type 2, a TGF-beta trap.
* The NHS-IL12 (M9241) immunocytokine is composed of 2 interleukin-12 (IL-12) heterodimers, each fused to one of the H-chains of the NHS76 antibody, which has affinity for both single- and double-stranded deoxyribonucleic acid (DNA). M9241 targets delivery of IL12, a proinflammatory cytokine that has been shown anti-tumor activity including objective responses in phase I clinical trials, to regions of tumor necrosis where DNA has become exposed, e.g., after radiation therapy.
* We hypothesize that released neo-epitopes upon increased DNA damage induced by radiation therapy together with the local proinflammatory action of M9241 will complement the anti-tumor activity of M7824 in locally advanced pancreas cancer.

Objectives:

* To determine the safety and tolerability and the recommended phase 2 dose (RP2D) of M7824 and M9241 in combination with stereotactic body radiotherapy (SBRT) as neoadjuvant/perioperative treatment in subjects with pancreas cancer.
* To determine a preliminary estimate of efficacy as best overall response (BOR) according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 of M7824 and M9241 in combination with SBRT as neoadjuvant/perioperative treatment in subjects with locally advanced pancreas cancer.

Eligibility:

* Histologically or cytologically proven pancreatic adenocarcinoma.
* Patient must be eligible to undergo stereotactic body radiation therapy (SBRT) (Cohorts 2-3).
* Patients must have measurable disease.
* Age greater than or equal to 18 years

Design:

* This is an open label Phase I/II trial. During phase I the safety and tolerability of M7824 and M9241 will be evaluated and recommended Phase II dose (RP2D) of M7824 and M9241 in combination with SBRT will be estimated. During phase II efficacy of the M7824 and M9241 in combination with SBRT will be examined.
* Patients will receive treatment in cycles consisting of 28 days (with exception of additional administer of M7824 alone in Phase IA).
* Treatment will continue until unacceptable toxicity or disease progression.
* If during treatment patient become candidate for curative surgery, treatment will be stopped and can be restarted after surgery in case if surgical exploration does not result in the successful removal of the tumor.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Histologically or cytologically proven pancreatic adenocarcinoma (subjects with endocrine or acinar pancreatic carcinoma are not eligible).
* Patients must have stage III or IV pancreatic cancer (Cohort 1) or locally advanced pancreas cancer (LAPC), either borderline resectable pancreas cancer or locally advanced, unresectable pancreas cancer (Cohorts 2 and 3).
* Patient must be eligible to undergo stereotactic body radiation therapy (SBRT) and have fiducial markers placed (any metal biliary stents are an acceptable alternative) (Cohorts 2-3).
* Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of bintrafusp alfa (M7824) and NHS-IL12 (M9241) in patients <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Must have measurable disease, per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* Adequate hematological function defined by:

  * white blood cell (WBC) count greater than or equal to 3 times 10^9/L
  * with absolute neutrophil count (ANC) greater than or equal to 1.0 times 10^9/L,
  * lymphocyte count greater than or equal to 0.5 times 10^9/L,
  * platelet count greater than or equal to 100 times 10^9/L, and
  * Hemoglobin (Hgb) greater than or equal to 9 g/dL (in absence of blood transfusion)
* Adequate renal function defined by:

  * Creatinine OR Measured or calculated creatinine clearance (CrCl) (estimated glomerular filtration rate (eGFR) may also be used in place of CrCl)

    * < 1.75 x institution upper limit of normal OR
    * greater than or equal to 45 mL/min/1.73 m^2 for participant with creatinine levels greater than or equal to 1.75 X institutional upper limit of normal (ULN)
  * Creatinine clearance (CrCl) or eGFR should be calculated per institutional standard
* Adequate hepatic function defined by:

  * a total bilirubin level less than or equal to 3 times ULN,
  * an aspartate aminotransferase (AST) level less than or equal to 5 times ULN,
  * alanine aminotransferase (ALT) level less than or equal to 5 times ULN
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression
* Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy.
* The effects of the study treatment on the developing human fetus are unknown; thus, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) at the study entry, for the duration of study treatment and up to 120 days after the last dose of the drug for males and up to 60 days for females. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Patient must be able to understand and willing to sign a written informed consent document.

EXCLUSION CRITERIA:

* Treatment with any investigational agent within 28 days before treatment initiation.
* Prior therapy with any antibody / drug targeting T cell coregulatory proteins (immune checkpoints) such as anti-Programmed cell death protein 1 (PD-1), anti-Programmed death-ligand 1 (PD-L1), or anti-cluster of differentiation 152 (CTLA-4) antibody.
* Anticancer treatment within designated period before treatment initiation including:

  * major surgical procedure (such as laparotomy) within 28 days
  * minor surgical procedure (such as biliary stenting) within 7 days
  * chemotherapy with published half-life known to be 72 hours within 7 days
  * chemotherapy with unpublished or half-life greater than 72 hours within 28 days
* Receipt of any organ transplantation, including allogeneic stem-cell transplantation, except of transplants that do not require immunosuppression (e.g., corneal transplant, hair transplant)
* Significant acute or chronic infections including tuberculosis (history of exposure or history of positive tuberculosis test; plus, presence of clinical symptoms, physical or radiographic findings)
* Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent with the exceptions:

  * diabetes type I, vitiligo, alopecia, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible;
  * subjects requiring hormone replacement with corticosteroids are eligible if the steroids are administered only for the purpose of hormonal replacement and at doses less than or equal to 10 mg of prednisone or equivalent per day;
  * administration of steroids for other conditions through a route known to result in a minimal systemic exposure (topical, intranasal, intro-ocular, or inhalation.
* Known severe hypersensitivity reactions to monoclonal antibodies (Grade greater than or equal to 3 National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) v5.0, any history of anaphylaxis or history of uncontrolled asthma.
* Known alcohol or drug abuse.
* Clinically significant cardiovascular / cerebrovascular disease as follows: cerebral vascular accident / stroke (< 6 months prior to treatment initiation), myocardial infarction (< 6 months prior to treatment initiation), unstable angina, congestive heart failure (New York Heart Association Classification Class greater than or equal to II), or serious cardiac arrhythmia.
* Administration of live vaccines within 30 days prior to treatment initiation.
* Human immunodeficiency virus (HIV), hepatitis C virus (HCV), hepatitis B virus (HBV) patients on antiviral drugs are excluded due to the absence of previous experience on combination of antiviral and this trial drugs and possible interaction.
* Subjects with a history of serious intercurrent chronic or acute illness, such as cardiac or pulmonary disease, hepatic disease, bleeding diathesis or recent (within 3 months) clinically significant bleeding events, or other illness considered by the Investigator as high risk for investigational drug treatment.
* Subjects unwilling to accept blood products as medically indicated.
* Female patients who are pregnant or breastfeeding. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with M7824 or M9241, breastfeeding should be discontinued.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2022-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Udo Rudloff, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. In addition, all large-scale genomic sequencing data will be shared with subscribers to database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Genomic data are available once genomic data are uploaded per protocol genomic data sharing (GDS) plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).
  Genomic data are made available via database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-C-0074.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 Phase 1A/Arm 1A Dose Level 0 De-Escalation: De-escalating doses of NHS-IL12 (M9241) in combination with bintrafusp alfa (M7824)
  M7824: Intravenous (IV) on Days 1 and 15 of every cycle
  M9241: Subcutaneous injection on Day 1 of every cycle
  M7824, 1200mg intravenous every 2 weeks; M9241, 16.8g/kg, subcutaneously, every 4 weeks
- Cohort 2 Phase 1B Arm 1B: No participants were enrolled on Cohort 2 Phase 1B Arm 1B. The study never progressed beyond stage 1A.
- Phase II Cohort 3 Arm 2: No participants were enrolled on Phase II Cohort 3 Arm 2. The study never progressed beyond stage 1A.
Period: Overall Study
Arm/Group | Cohort 1 Phase 1A/Arm 1A Dose Level 0 De-Escalation | Cohort 2 Phase 1B Arm 1B | Phase II Cohort 3 Arm 2
Started | 3 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 3 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0
Not completed — Death | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cohort 1 Phase 1A/Arm 1A Dose Level 0 De-Escalation
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (10.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase 2 Dose (RP2D) of NHS-IL12 (M9241) Given With Bintrafusp Alfa (M7824) in Combination With Stereotactic Body Radiation Therapy (SBRT) as Neoadjuvant / Perioperative Treatment in Participants With Pancreas Cancer
Description: The recommended phase 2 dose (RP2D) is the dose level of M9241 in combination with M7824 at which ≤1 of 6 individuals experienced a dose limiting toxicity (DLT) during the first cycle (28 days) of combinational treatment with M9241 and M7824. A DLT is any Grade ≥ 3 adverse events occurring during the first 28 days of treatment except adverse events unrelated, or unlikely related to study agents and probably or definitely related to other causes.
Time Frame: First 28 days of treatment
Population: Data was not collected because the study never got beyond phase 1A and was terminated, thus the RP2D was not found.
Arm/Group | Cohort 1 Phase 1A/Arm 1A Dose Level 0 De-Escalation
Number analyzed (Participants) | 0

2. Primary Outcome: Number of Participants With ≥Grade 3 Toxicities Possibly, Probably, or Definitely Related to Treatment of Bintrafusp Alfa (M7824) and NHS-IL12 (M9241) in Combination With Stereotactic Body Radiation Therapy (SBRT)
Description: Adverse events were assessed using the Common Terminology Criteria for Adverse Events (CTCAE)v5.0. Grade 3 is severe, Grade 4 is life-threatening, and Grade 5 is death related to adverse events.
Time Frame: Date treatment consent signed to date off study, approximately 4 months and 13 days.
Population: No data were collected because no participants received SBRT WITH M7824 and M9241.
Arm/Group | Cohort 1 Phase 1A/Arm 1A Dose Level 0 De-Escalation
Number analyzed (Participants) | 0

3. Primary Outcome: Best Overall Response (BOR) According to the Response Evaluation Criteria in Solid Tumors (RECIST) of Bintrafusp Alfa (M7824) & NHS-IL12 (M9241) in Combination With Stereotactic Body Radiation Therapy in Participants With Locally Advanced Pancreas Cancer
Description: Best overall response is measured from the time measurement criteria are met for complete response or partial response until the first date that recurrent or progressive disease is objectively documented using the Response Evaluation Criteria in Solid Tumors (RECIST). Complete Response (CR) is disappearance of all target lesions. Partial Response (PR) is at least a 30% decrease in target lesions. In the case of a PR or CR a confirmatory computed tomography or magnetic resonance imaging scan should be done no sooner than 4 weeks. Progressive Disease (PD) is at least a 20% increase in target lesions and/or the appearance of new lesions.
Time Frame: time measurement criteria are met for complete response or partial response until the first date that recurrent or progressive disease is objectively documented
Population: No data were collected because no participants received SBRT WITH M7824 and M9241.
Arm/Group | Cohort 1 Phase 1A/Arm 1A Dose Level 0 De-Escalation
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Survival (OS) in Participants After Completion of Radiation Therapy (RT) in Combination With NHS-IL12 (M9241) and Bintrafusp Alfa (M7824)
Description: Overall survival is defined as date of on-study to the date of death from any cause or last follow up.
Time Frame: date of on-study to the date of death from any cause or last follow
Population: Data were not collected because no participants received RT.
Arm/Group | Cohort 1 Phase 1A/Arm 1A Dose Level 0 De-Escalation
Number analyzed (Participants) | 0

5. Secondary Outcome: Progression-free Survival (PFS) for All Participants
Description: Progression free survival is defined as the time interval from start of treatment to documented evidence of disease progression. Progression was measured using the Response Evaluation Criteria in Solid Tumors (RECIST) and is at least a 20% increase in target lesions and/or the appearance of new lesions.
Time Frame: Time interval from start to treatment to disease progression, an average of 4 months.
Population: 2/3 participants were evaluable because one participant did not make it to his first restaging scan.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 Phase 1A/Arm 1A Dose Level 0 De-Escalation
Number analyzed (Participants) | 2
Months | 4 [2.3 to 5.9]

6. Secondary Outcome: Progression-free Survival (PFS) for Participants Who Did Not Undergo Surgical Resection
Description: as for outcome 5
Time Frame: time interval from start of treatment to documented evidence of disease progression
Population: 2/3 participants were evaluable because one participant did not make it to his first restaging scan.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 Phase 1A/Arm 1A Dose Level 0 De-Escalation
Number analyzed (Participants) | 2
Months | 4 [2.3 to 5.9]

7. Secondary Outcome: Fraction of Participants With Locally Advanced, Non-metastatic Pancreas Cancer (LAPC) Who Are Able to Undergo Surgical Resection After Bintrafusp Alfa (M7824) and NHS-IL12 (M9241) in Combination With Stereotactic Body Radiation Therapy (SBRT) Treatment
Description: Fraction of participants with LAPC who are able to undergo surgical resection after M7824, M9241 and SBRT.
Time Frame: At time of surgical resection
Population: No data were collected because no participants had M7824 and M9241 WITH SBRT.
Arm/Group | Cohort 1 Phase 1A/Arm 1A Dose Level 0 De-Escalation
Number analyzed (Participants) | 0

8. Secondary Outcome: Time-to-recurrence of the Disease For Participants Who Underwent Surgical Resection After Bintrafusp Alfa (M7824) and NHS-IL12 (M9241) in Combination With Stereotactic Body Radiation Therapy (SBRT) Treatment
Description: Time-to-recurrence of disease is defined as time from surgical resection to disease recurrence (expressed in months).
Time Frame: At disease recurrence after surgical resection
Population: No participants made it to surgical resection nor had SBRT.
Arm/Group | Cohort 1 Phase 1A/Arm 1A Dose Level 0 De-Escalation
Number analyzed (Participants) | 0

9. Secondary Outcome: Complete Pathological Response Rate(s) For Participants Who Underwent Surgical Resection After Bintrafusp Alfa (M7824) and NHS-IL12 (M9241) in Combination With Stereotactic Body Radiation Therapy (SBRT) Treatment
Description: Complete Pathological Response is defined as the fraction of participants who had a complete pathologic response of all participants who underwent surgery. Complete pathological response was measured using the Response Evaluation Criteria in Solid Tumors and is defined as
Time Frame: At time of surgical resection
Population: No data were collected because no participants received M7824, M9241 WITH SBRT.
Arm/Group | Cohort 1 Phase 1A/Arm 1A Dose Level 0 De-Escalation
Number analyzed (Participants) | 0

10. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0).
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 4 months and 13 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Phase 1A/Arm 1A Dose Level 0 De-Escalation
Number analyzed (Participants) | 3
Participants | 3

11. Other Pre Specified Outcome: Number of Participants With a Dose-limiting Toxicity (DLT)
Description: A DLT is any Grade ≥ 3 adverse events occurring during the first 28 days of treatment except adverse events unrelated, or unlikely related to study agents and probably or definitely related to other causes.
Time Frame: First 28 days of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Phase 1A/Arm 1A Dose Level 0 De-Escalation
Number analyzed (Participants) | 3
Participants | 1

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 4 months and 13 days.
Arm/Group | Cohort 1 Phase 1A/Arm 1A Dose Level 0 De-Escalation
All-Cause Mortality (participants affected / at risk) | 1/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 Phase 1A/Arm 1A Dose Level 0 De-Escalation (N=3)
Anemia (Blood and lymphatic system disorders) | 1 (2)
Vascular disorders - Other, gastrointestinal hemorrhage (Vascular disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 Phase 1A/Arm 1A Dose Level 0 De-Escalation (N=3)
Anemia (Blood and lymphatic system disorders) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood and lymphatic system disorders - Other, elevated white blood cells (Blood and lymphatic system disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 1 (3)
Hypotension (Vascular disorders) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (4)
Malaise (General disorders) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, rash (Skin and subcutaneous tissue disorders) | 1 (1)
Thrush (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-10): https://cdn.clinicaltrials.gov/large-docs/86/NCT04327986/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-08): https://cdn.clinicaltrials.gov/large-docs/86/NCT04327986/ICF_001.pdf